CLINICAL TRIAL: NCT04455035
Title: DynaCleft® Effects on Soft Tissues and on Quality of Life for Incomplete Unilateral Cleft Lip Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Brett Thomas Chiquet, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-DB-20-0311
Record Dates: First submitted 2020-06-26; First posted 2020-07-02 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Cleft Lip and Palate
Keywords: Dynacleft
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Retrospective Group(Control) (Active Comparator)
  Interventions: Other: Comparator: Retrospective Group(Control)
- Prospective Group (Experimental)
  Interventions: Device: Prospective Group

INTERVENTIONS:
Other: Comparator: Retrospective Group(Control) — The control group for this study will be obtained from a retrospective chart review of electronic health records of patients with incomplete cleft lip who underwent surgery without any presurgical interventions.
  Arms: Retrospective Group(Control)
Device: Prospective Group — The study population for the prospective aspect will include recruited newborns with untreated unilateral incomplete cleft lip.
  DynaCleft® + Nasal Elevator therapy will be discussed with parent(s) as a presurgical orthopedic option while awaiting primary cleft lip surgical repair that typically occurs between the ages of 3 to 6 months.Study duration will be up to three months of presurgical intervention.Photographs are to be taken at initial visit prior to presurgical intervention and later at completion of the DynaCleft® therapy immediately prior to lip surgery. Angles to be pictured are to include the standard anterior-posterior, profile, and worms-eye view.
  Linear measurements will be obtained with a ruler and registered in millimeters. A goniometer will be used to measure angles.
  Arms: Prospective Group

SUMMARY:
The purpose of this study is to examine the effectiveness of the DynaCleft® system on soft tissues of infants with unilateral incomplete cleft lip and to assess influences on quality of life for infants who underwent DynaCleft® and that of their families.

ELIGIBILITY:
Inclusion Criteria:

Retrospective Group:

* Unilateral cleft lip with or without cleft palate
* Patients of a single surgeon (Matthew Greives, MD)
* Patients with complete photographs:

  * After birth, first visit
  * At cleft lip repair (3-4 months)
  * Post-operative cleft repair (about 1 year of age)

Prospective Group:

* Patients with incomplete unilateral cleft lip with or without cleft palate
* Patients of any surgeon

Exclusion Criteria:

Retrospective Group:

* Bilateral cleft lip or complete unilateral cleft lip
* Patients operated on by other primary surgeons
* Patients with incomplete photo records will be evaluated to determine if the patient should be excluded

Prospective Group:

* Patients with bilateral cleft lip or complete unilateral cleft lip
* Patients whose parents refuse to consent to inclusion
* Patients with tape allergies to the adhesive of the DynaCleft®
* Patients with syndromic craniofacial conditions or Tessier type facial clefts

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett T Chiquet, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Retrospective Group(Control) | Prospective Group
Started | 20 | 4
Completed | 20 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retrospective Group(Control) | Prospective Group | Total
Number analyzed (Participants) | 20 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 4 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data for this measure were not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Changes in Soft Tissue as Indicated by Width of the Cleft Lip Measured From Extraoral Clinical Photographs
Description: Width of the cleft lip was measured from extraoral clinical photographs. Data reported is width of cleft lip at 3 months minus width of cleft lip at time of initial examination.
Time Frame: initial time of examination with study team, time of surgery (3 months post intervention)
Measure: Mean (Standard Deviation); unit: pixels
Arm/Group | Retrospective Group(Control) | Prospective Group
Number analyzed (Participants) | 20 | 4
pixels | 0.601 (0.236) | 0.435 (0.111)
Statistical Analysis 1: Comparison: Retrospective Group(Control) vs Prospective Group; Test type: Other — ttest; p = 0.0088, t-test, 2 sided

2. Primary Outcome: Changes in Soft Tissue as Indicated by Columellar Angle Measured From Extraoral Clinical Photographs
Description: Columellar angle was measured from extraoral clinical photographs. Data reported is columellar angle at 3 months minus columellar angle at time of initial examination.
Time Frame: initial time of examination with study team, time of surgery (3 months post intervention)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Retrospective Group(Control) | Prospective Group
Number analyzed (Participants) | 20 | 4
degrees | 54.93 (5.124) | 64.75 (4.991)
Statistical Analysis 1: Comparison: Retrospective Group(Control) vs Prospective Group; Test type: Other — ttest; p = 0.00001, t-test, 2 sided

3. Primary Outcome: Changes in Soft Tissue as Indicated by Nostril Height Measured From Extraoral Clinical Photographs
Description: Data was not collected for this outcome. Data was not collected for this outcome. Data was not collected for this outcome. Data was not collected for this outcome. Data was not collected for this outcome.
Time Frame: initial time of examination with study team, time of surgery (3 months post intervention)
Population: Data was not collected for this outcome measure.
Arm/Group | Retrospective Group(Control) | Prospective Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Changes in Soft Tissue as Indicated by Nostril Width Measured From Extraoral Clinical Photographs
Description: as for outcome 3
Time Frame: initial time of examination with study team, time of surgery (3 months post intervention)
Population: Data was not collected for this outcome measure.
Arm/Group | Retrospective Group(Control) | Prospective Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Average Number of Responses Indicating Improvement, no Change, or Decrease in Quality of Life as Assessed by the Infant and New Parent Quality of Life Questionnaire
Description: The Infant and New Parent Quality of Life questionnaire consists of 22 questions related to quality of life. For each question, it was determined whether the response at 3 months indicated an improvement, no change, or a decrease in quality of life relative to the response at the time of initial examination. The average number with an improvement in quality of life (averaged over all 22 questions), the average number who had no change in quality of life (averaged over all 22 questions), and the average number who had a decrease in quality of life (averaged over all 22 questions) are reported.
Time Frame: initial time of examination with study team, time of surgery (3 months post intervention)
Population: Data for this outcome measure were not collected from the retrospective arm, as IRB approval was not requested to contact retrospective participants.
Measure: Mean (Standard Deviation); unit: number of responses
Arm/Group | Retrospective Group(Control) | Prospective Group
Number analyzed (Participants) | 0 | 4
number of responses
  improvement in quality of life |  | 2.27 (0.83)
  no change in quality of life |  | 1.68 (0.84)
  decrease in quality of life |  | 0 (0)

ADVERSE EVENTS:
Time Frame: 4 months
Description: Parents of patients in "treatment"/prospective arm could report challenges/pitfalls to investigator team, and investigator team met with family monthly (4 months, 20-30 minute appointments) to collect data and evaluate. Adverse event data were not collected for the retrospective arm, as IRB approval was not requested to contact retrospective participants.
Arm/Group | Retrospective Group(Control) | Prospective Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 0/0 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT04455035/Prot_SAP_000.pdf